CLINICAL TRIAL: NCT03679741
Title: Initial Evaluation of Investigational Lenses Manufactured on a New Production Line
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6283
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL/CONTROL (Experimental): Subjects that are 18 to 49 years of age and current spherical soft contact lens wears will be randomized into one of two lens wear sequences. Subjects will wear the Test and Control lenses for two weeks each with one of the study lenses being worn twice for a total of 6 weeks.
  Interventions: Device: CONTROL Lens; Device: TEST Lens
- CONTROL/TEST/TEST (Experimental): Subjects that are 18 to 49 years of age and current spherical soft contact lens wears will be randomized into one of two lens wear sequences. Subjects will wear the Test and Control lenses for two weeks each with one of the study lenses being worn twice for a total of 6 weeks.
  Interventions: Device: CONTROL Lens; Device: TEST Lens

INTERVENTIONS:
Device: CONTROL Lens — Acuvue OASYS
Device: TEST Lens — senofilcon A

SUMMARY:
This study is a randomized, 4-visit, subject-masked, 2x3 bilateral crossover, dispensing trial. Each study lens will be worn bilaterally in a daily wear (DW) modality for at least 6 hours per day and 5 days per week for approximately two weeks each. The subject will wear either the Test or Control lens twice and the other study lens once.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read and sign the Informed Consent form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Healthy adult males or females age ≥18 and ≤49 years of age with signed informed consent. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them.
4. The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and -6.00 D.
5. The subject's refractive cylinder must be ≤ 1.00 D in each eye.
6. The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
7. Subjects must own a wearable pair of spectacles.
8. The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of DW per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis.
9. Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week.
10. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
3. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral (e.g., Chlor-Trimeton, and Benadryl) and ophthalmic antihistamines, oral phenothiazines (e.g., Haldol, Mellaril, Thorazine, Elavil, Pamelor, Compazine), oral and ophthalmic Beta-adrenergic blockers (e.g., Propranolol, Timolol, and Practolol), systemic steroids, and any prescribed or over the counter (OTC) ocular medication.
4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion.
5. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), LASIK, etc.).
6. Any Grade 3 or greater slit lamp findings (e.g.., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
7. Any known hypersensitivity or allergic reaction to Optifree® PureMoist® multi-purpose care solution or Eye-Cept® rewetting drop solution.
8. Any ocular infection, allergy or clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca, ocular hypertension), or ocular conditions (e.g. strabismus), which might interfere with the study.
9. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
10. Toric, extended wear, monovision or multi-focal contact lens correction.
11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
12. Participation in clinical trials involving the Test lens within 3 months prior to study enrollment.
13. History of binocular vision abnormality or strabismus.
14. Employee, relative or friends of employees of any ophthalmic company, or investigational clinic (e.g., Investigator, Coordinator, Technician).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Randall Go, OD, San Francisco, California
  - VRC-East, Jacksonville, Florida
  - Sacco Eye Group, Vestal, New York
  - Pickens Eye Care, Pickens, South Carolina
  - William J. Bogus, OD, FAAO, Salt Lake City, Utah
  - Botetourt Eyecare, LLC, Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 126 subjects were enrolled into this study. Of those enrolled, 120 subjects were randomized and dispensed at least one study lens. Of the dispensed subjects, 110 completed the study, while 10 subjects were discontinued.
Groups:
- Test/Control/Control: Subjects that were randomized to receive the test lens during the first period and the control lens during both the second and third periods.
- Control/Test/Test: Subjects that were randomized to receive the control lens during the first period and the test lens during both the second and third periods.
Period: Period 1
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 59 | 61
Completed | 57 | 58
Not Completed | 2 | 3
Not completed — No longer meet eligibility criteria | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 57 | 58
Completed | 54 | 56
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Period 3
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 54 | 56
Completed | 54 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Dispensed Subjects: All subjects dispensed at least one study lens regardless of randomization.
Arm/Group | All Dispensed Subjects
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.3 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 11
  Black or African American | 7
  White | 102
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort Score
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Test: Subjects that wore the Test lens during any of the three periods during the study.
- Control: Subjects that wore the Control lens during any of the three periods during the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 109 | 109
Units on a Scale | 59.30 (23.779) | 58.54 (22.303)
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 30 participants randomized in a 1:1 fashion between the two lens wear sequences would have at least 80% power to detect a 5 point difference between the test and control lenses with respect to overall comfort at the 2-week follow-up. Sample size was determined using Stroup's Method (alpha=0.05); Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE scores; Bayesian multivariate normal random-effe; A 95% Credible Interval for the Posterior mean difference between the Test and Control was used to test for non-inferiority; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-1.9 to 5.8], Standard Deviation 1.99 — Mean difference was calculated as test minus control

2. Primary Outcome: Vision Satisfaction in Bright Lighting
Description: Vision satisfaction in bright light was assessed using the individual item" I was satisfied with the quality of my vision in bright lighting" from the CLUE™ questionnaire. This item used the response scale, 1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree and 5: Strongly Agree. CLUE is the Contact Lens User Experience™ questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. The Proportion of responses in each category were reported for each lens type.
Time Frame: 2-Week Follow-up
Population: subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Proportion of participants
Arm/Group | Test | Control
Number analyzed (Participants) | 109 | 109
Proportion of participants
  Strongly Agree | 0.22 | 0.11
  Agree | 0.622 | 0.583
  Neither Agree Nor Agree | 0.098 | 0.141
  Disagree | 0.061 | 0.135
  Strongly Disagree | 0.00 | 0.031
Statistical Analysis 1: Comparison: Test vs Control; Test type: Non-Inferiority — A cumulative odds ratio non-inferiority margin of 0.67 was used. This margin is based on no more than a 10% difference in proportion between the Test and the Control lenses. The odds ratio represents the cumulative odds ratio of having a higher rating/experience of the Test lens compared to the Control lens; Bayesian multinomial random-effects mode; A 95% Credible Interval for the odds ratio, was used to test for non-inferiority; Odds Ratio (OR) = 3.97, 95% CI 2-sided [2.27 to 6.62], Standard Deviation 1.138 — Odds ratio was calculated as test over control

3. Primary Outcome: Distance Monocular LogMAR Visual Acuity
Description: Distance Monocular LogMAR visual acuity was assessed at 4 meters using an ETDRS chart under high illumination low contrast (room illumination > 400 lux and chart luminance 120-200 cd/m2) and low illumination high contrast (room illumination <2.5 lux and chart luminance 2.0 - 5.0 cd/m2 at the 2-week follow-up for each subject eye. The average visual acuity for each lens was reported.
Time Frame: 2-Week Follow-up
Population: subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 109 | 109
Number analyzed (Eyes) | 218 | 218
logMAR
  High Illumination low contrast | 0.10 (0.086) | 0.14 (0.089)
  Low illumination high contrast | 0.06 (0.082) | 0.08 (0.085)
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 4 participants randomized in a 1:1 fashion between the two lens types would have at least 80% power to detect non-inferiority with respect to visual acuity (logMAR) at the 2-week follow-up. Sample size was determined using Stroup's method. The analysis presented below, summarizes the low luminance high contrast lighting condition; Test type: Non-Inferiority — A non-inferiority margin of 0.05 logMAR was used. This margin corresponds to a half line difference. Non-inferiority was declared if the upper bound of the 95% credible interval was below 0.05 logMAR; Bayesian multivariate normal model; with random effects; Mean Difference (Final Values) = -0.022, 95% CI 2-sided [-0.037 to -0.008], Standard Deviation 0.0074 — Mean difference was calculated as Test minus Control
Statistical Analysis 2: Comparison: Test vs Control; It was calculated that 4 participants randomized in a 1:1 fashion between the two lens types would have at least 80% power to detect non-inferiority with respect to visual acuity (logMAR) at the 2-week follow-up. Sample size was determined using Stroup's method. The analysis presented below, summarizes the high illumination low contrast lighting condition; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Bayesian multivariate normal model; with random effect; Mean Difference (Final Values) = -0.034, 95% CI 2-sided [-0.049 to -0.020], Standard Deviation 0.0075 — Mean difference was calculated as Test minus Control

4. Primary Outcome: Contact Lens Fitting Acceptance Rate
Description: Contact lens fitting acceptance was assessed for each subject eye using a biomicroscope at all study visits. Lens fit was a binary variable where acceptable lens fit=1 and unacceptable lens fit=0. The percentage of eyes with acceptable lens fit was reported for each lens.
Time Frame: Up to 2-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 109 | 109
Number analyzed (eyes) | 218 | 218
percentage of eyes | 100 | 100
Statistical Analysis 1: Comparison: Test; It was calculated that 65 participants were required to show that the acceptable lens fitting for the Test lens would be superior to 90% with at least 80% power. Sample size was determined using simulations methods for repeated measures; Test type: Superiority — A superiority margin of 90% was used. Superiority was concluded if the lower limit of the 95% credible interval was above 90%; Bayesian beta- binomial model; for correlated binary data; Mean Percentage of eyes = 100.0, 95% CI 2-sided [99.0 to 100.0], Standard Deviation 0.002

5. Primary Outcome: Number of Grade 3 or Higher Slit Lamp Findings
Description: Slit Lamp Findings (SLF) were assessed using a biomicroscope and was graded using the FDA grading scale (Grade: 0, 1,2, 3 and 4) with grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e. Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe). This was performed on each subject eye at every study visit (baseline, unscheduled visits and 2-week follow-up). The data was then dichotomized into two groups. Those with grade 3 or higher and those with grade 2 or lower. The proportion of eyes with SLF with grade 3 or higher by lens was reported.
Time Frame: Up to 2-Week Follow-up
Population: All subjects dispensed a study lens.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 109 | 109
Number analyzed (eyes) | 218 | 218
proportion of eyes | 0.005 | 0.000
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 50 participants randomized in a 1:1 fashion between the two lens wear sequences would have at least 80% power to detect 5% difference between the Test and Control lens with respect to the proportion of eyes with Grade 3 or higher slit lamp findings across all study visits. Sample size was determined using simulations methods; Test type: Non-Inferiority — A non-inferiority cumulative odds ratio margin of 2 was used. This margin corresponds to no more than a 5% difference between the Test and Control lenses assuming the Control reference rate does not exceed 5%. Non-inferiority was declared if the upper bound of the 95% credible interval was below 2; Bayesian beta-binomial hierarchical; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-0.004 to 0.008], Standard Deviation 0.003 — Mean difference was calculated as Test minus Control

6. Secondary Outcome: Overall Quality of Vision Score
Description: Overall quality of vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test | Control
Number analyzed (Participants) | 109 | 109
Units on a Scale | 62.25 (18.460) | 58.47 (18.707)
Statistical Analysis 1: Comparison: Test vs Control; Sample size was based on primary endpoints only; Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE scores; Bayesian multivariate normal model; for random effects; Mean Difference (Final Values) = 5.6, 95% CI 2-sided [3.1 to 8.1], Standard Deviation 1.29 — Mean difference was calculated as test minus control

7. Secondary Outcome: Overall Handling Scores
Description: Overall handling was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Test | Control
Number analyzed (Participants) | 109 | 109
Units on a Scale | 66.24 (19.185) | 64.66 (20.460)
Statistical Analysis 1: Comparison: Test vs Control; Sample size was based on primary endpoints only; Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE scores; Bayesian multivariate normal model; for random effects; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-0.6 to 5.5], Standard Deviation 1.56 — Mean difference was calculated as test minus control

8. Secondary Outcome: Overall Quality of Vision Indoors
Description: Overall Quality of Vision Indoors was assessed using the individual item" Overall Quality of Vision Indoors" from questionnaire assessing contact lens performance. This item used the response scale, 0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor. The Proportion of responses in each category were reported for each lens type.
Time Frame: 2-Week Follow-up
Population: subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Proportion of participants
Arm/Group | Test | Control
Number analyzed (Participants) | 109 | 109
Proportion of participants
  Excellent | 0.433 | 0.374
  Very Good | 0.396 | 0.393
  Good | 0.128 | 0.184
  Fair | 0.043 | 0.049
  Poor | 0 | 0
  Not Applicable | 0 | 0
Statistical Analysis 1: Comparison: Test vs Control; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Bayesian multinomial random-effects; A 95% Credible Interval for the odds ratio, was used to test for non-inferiority; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.00 to 2.82], Standard Deviation 0.459 — Odds ratio was calculated as test over control

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 6-Weeks per subject.
Groups:
- Test: Subjects that wore the Test lens during any of the 3 period during the study.
- Control: Subjects that wore the Controllens during any of the 3 period during the study.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03679741/SAP_000.pdf
  • Study Protocol (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT03679741/Prot_001.pdf